CLINICAL TRIAL: NCT04492592
Title: The J(Amaican and) U(Nited) S(Tates) Media? Programme: A Food-Focused Media Literacy Intervention for Americanized Adolescents and Mothers Globally
Brief Title: JUS Media? Programme: A Food-Focused Media Literacy Intervention for Americanized Adolescents and Mothers Globally
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: The University of The West Indies (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Gail Marcia Ferguson, Associate Professor, University of Minnesota
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 17182
Record Dates: First submitted 2019-08-15; First posted 2020-07-30 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Nutrition Poor
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not told what arm of the intervention they were in (i.e., they were not told if they were receiving the intervention or not).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Workshop Only (Experimental): 2 session weekend face:face workshop for adolescent-mother pairs
  Interventions: Behavioral: SMS/Texting
- Workshop + SMS/Texting (Experimental): 2 session weekend face:face workshop for adolescent-mother pairs followed by 8 weeks of supplementary text messages (NOTE: there was no 'SMS/texting-only' arm of this study)
  Interventions: Behavioral: Workshop; Behavioral: SMS/Texting
- Control (No Intervention): No intervention provided.

INTERVENTIONS:
Behavioral: Workshop — Workshop
  Arms: Workshop + SMS/Texting
Behavioral: SMS/Texting — SMS/Texting
  Arms: Workshop + SMS/Texting; Workshop Only

SUMMARY:
The J(amaican and) U(nited) S(tates) Media? Programme is a culturally-tailored food-focused media literacy preventive intervention designed to promote healthier eating habits among remotely acculturating early adolescents and their mothers in Jamaica (i.e., they have internalized American culture) and are exposed to U.S. food advertising. The JUS Media? Programme consists of a 2-session face:face weekend workshop for adolescent-mother pairs supplemented by 8 weeks of SMS/text messages to reinforce workshop themes. Adolescents and their mothers learn critical thinking skills to combat the unhealthy food messages they encounter in food advertising, particularly advertising on U.S. cable TV. The efficacy of the JUS Media? Programme was evaluated with a small experimental study utilizing a randomized controlled trial design among adolescents and mothers in Jamaica.

DETAILED DESCRIPTION:
The Western diet is common in the United States and has a lot of salt, sugar, and fat. Modern globalization has shifted eating habits in many countries toward this unhealthy Western diet. For example, U.S. cable TV in other countries promotes this Western diet through advertisements for junk foods and sugary drinks. This is a major concern because experimental research studies show that seeing food advertising while watching TV leads to eating more food afterwards. Research studies also show that people who watch a lot of TV tend to think that junk food is not that harmful.

Researchers now believe that some people living outside the U.S. are drawn to the U.S. culture and lifestyle and can become "Americanized" through a process called remote acculturation. These Americanized people in other countries such as Jamaica are mostly teenagers, but sometimes also adults. Americanized people outside the United States are even more likely to adopt the unhealthy Western diet even though they have never lived in the United States. In research the investigators did before getting this grant, they showed that Americanized youth and mothers in Jamaica watched more hours of U.S. cable daily and also ate more unhealthy food. This led them to develop a new healthy eating education program for Americanized families in Jamaica that highlighted the role of U.S. media - the "J(amaican) U(nited) S(tates) Media? Programme". The JUS Media? Programme teaches young people and mothers to question the health messages in food advertising on U.S. cable TV so that they can be smarter and healthier consumers. For example, the JUS Media? Programme covers the recommended food guidelines in Jamaica and teaches adolescents and their mothers the principles of media literacy, such as to think about "who is the source of this message?" "what do they want you to do?" and "what information is missing?". Finally, the JUS Media? Programme teaches participants to use these media literacy principles to challenge unhealthy food advertisements by creating smart, funny parody versions called subvertisements.

In this project,the investigators evaluated how well the JUS Media? Programme worked for 7th graders and their mothers in Jamaica. About 30 adolescents and their mothers got a 2-session workshop, another 30 families got the workshop and text messages, and another 30 families did not get any part of the program.

ELIGIBILITY:
Inclusion criteria:

• 7th grader enrolled in the participating schools and present at school on the days of recruitment.

Exclusion criteria for each adolescent or mother seeking to enroll:

* mother/student was not born in Jamaica
* mother/student is not a Jamaican citizen
* mother/student is a citizen (including dual citizen) of the United States
* mother/student has not lived in Jamaica for the past 15 years (mother) or 8 years (student)
* mother and student do not live together
* mother has been primary guardian for <5 years
* study screening scores show no U.S. TV usage or no affinity for the U.S. culture, and very low junk food consumption

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Dietary Intake Using a 24-Hour Recall Method | 4 measurement points: baseline, 4 weeks, 6 weeks, 17-20 weeks (study ended at this final timepoint).
  24-Hour Recall. Each participant reported detailed information on all foods and beverages consumed in the previous 24 hours via structured interviews with open-ended responses over the phone, and reported dietary intake was coded into coded for the presence (1) or absence (0) of fruits, raw vegetables, cooked vegetables, fats/oils, and sugary foods/beverages (aligning with the major national food groups of the population studied).
CHANGE IN STAGE OF CHANGE TOWARDS HEALTHY EATING | 4 measurement points: baseline, 4 weeks, 6 weeks, 17-20 weeks (study ended at this final timepoint).
  A stages of change measure of healthy eating (Wright et al., 2015) was adapted to measure participants' adherence to 5 additional food-based dietary guidelines of the Jamaica Ministry of Health. Participants reported their adherence to each dietary guideline using a 1-6 likert type scale ranging from 1 "precontemplation stage (No, and I do not intend to [insert wording from guideline]...in the next 6 months" to 6 "total abstinence (I do not consume...[insert wording from guideline)." Higher scores on this scale represent being closer to one's healthy eating goal.

SECONDARY OUTCOMES:
CHANGE IN FOOD-FOCUSED MEDIA LITERACY | 4 measurement points: baseline, 4 weeks, 6 weeks, 17-20 weeks (study ended at this final timepoint).
  Food-focused media literacy was measured with a 14-item scale (Powell & Gross, 2018). Participants responded on a 4-point likert type scale ranging from 1 (strongly disagree) to 4 (strongly agree). Higher scores on this scale represent higher food-focused media literacy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferguson GM, Meeks Gardner JM, Nelson MR, Giray C, Sundaram H, Fiese BH, Koester B, Tran SP, Powell R. Food-Focused Media Literacy for Remotely Acculturating Adolescents and Mothers: A Randomized Controlled Trial of the "JUS Media? Programme". J Adolesc Health. 2021 Dec;69(6):1013-1023. doi: 10.1016/j.jadohealth.2021.06.006. Epub 2021 Jul 17. PMID 34281754